CLINICAL TRIAL: NCT00047827
Title: A Phase 2, Open-Label, Non-Comparative Trial of Micafungin (FK463) in Combination With Liposomal Amphotericin B (AmBisome) as First-Line Therapy in the Treatment of Invasive Aspergillosis
Brief Title: Trial of Micafungin (FK463) in Combination With Liposomal Amphotericin B (AmBisome) for Aspergillosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-0-125; FG463-21-11
Record Dates: First submitted 2002-10-18; First posted 2002-10-24 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Aspergillosis
Keywords: Aspergillus; Aspergillosis; Anti-Fungal; AmBisome; Micafungin
MeSH Terms: conditions — Aspergillosis | interventions — Micafungin; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Micafungin; Drug: Liposomal Amphotericin B

INTERVENTIONS:
Drug: Micafungin — IV
  Other Names: Mycamine; FK463
Drug: Liposomal Amphotericin B — IV
  Other Names: AmBisome

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of micafungin in combination with AmBisome as first-line therapy in the treatment of invasive aspergillosis.

ELIGIBILITY:
Inclusion Criteria

* Have proven or probable systemic infection with Aspergillus species and have received no more than 96 hours of prior therapeutic doses of systemic antifungal therapy

Exclusion Criteria

* Has abnormal liver test parameters, e.g., AST or ALT > 10 times upper limit of normal
* Has allergic bronchopulmonary aspergillosis, aspergillomas, or with sinus aspergillosis or external otitis who do not have evidence of tissue invasion
* Has life expectancy of less than five days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2002-12; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment response defined as complete or partial response | Day 28, end of combined therapy and Day 84

SECONDARY OUTCOMES:
Clinical Response | Day 28, end of combined therapy and Day 84
Radiological Response | Day 28, end of combined therapy and Day 84
Mycological Response | Day 28, end of combined therapy and Day 84
Survival at Day 84 | Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (7):
- United States (7):
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - St Louis, Missouri
  - Memphis, Tennessee
  - Houston, Texas